CLINICAL TRIAL: NCT03144791
Title: Lnfluence of Light Conditions on Brain Activity, Response Time, Autonomic Nervous Response, and Emotion in the Elderly and Young Adults
Brief Title: Lighting and Human Response in Motor Time, Autonomic Nervous System, and Emotion
Acronym: LiHR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/092.L006
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Physical Activity; Emotions; Autonomic Nervous System Imbalance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- elderly , young adults: Participants are in 9 light conditions, 5 minute for each condition.

SUMMARY:
Light influences on human movement, autonomic nervous system, and emotion. It is inconclusive whether illuminance (Ev) and colour temperature (Tc) is appropriate to human movement, autonomic nervous systme, and emotion. Effect of Ev and Tc on responses of movement, autonomic nervous system, and emotion in human is investigated.

DETAILED DESCRIPTION:
The adult and elderly sign informed consent form. They sit in a room where Ev and Tc is adjusted. During sitting they are measured response of movement, autonomic nervous system, and emotion.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 79 years old
* Normal visual acuity with or without own glasses or contact lens
* Normal visual field
* Normal visual color perception
* Able to following commands
* Able to read, write, and understand in Thai language
* Able to sit independently with or without support
* Able to move dominant upper limb
* No pain in dominant Shoulder, Elbow, Wrist, and Hand during movement

Exclusion Criteria:

* Aggravated pain at trunk and lower limb during movement of dominant upper limb
* Having Neurological disorders
* Having uncontrolled diseases
* Having psychological problems

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
motor response time | 1 minute
  ms

SECONDARY OUTCOMES:
Brain activity | 5 minutes
  microvolt
Heart rate variability | 2 minutes
  millisecond
emotion | 2 minutes
  score
skin conductance level | 2 minute
  microsiemens

CONTACTS AND LOCATIONS:
Overall Officials: Vimonwan Hiengkaew, PhD, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuijsters A, Redi J, de Ruyter B, Heynderickx I. Lighting to Make You Feel Better: Improving the Mood of Elderly People with Affective Ambiences. PLoS One. 2015 Jul 20;10(7):e0132732. doi: 10.1371/journal.pone.0132732. eCollection 2015. PMID 26192281
- [Background] Hanford N, Figueiro M. Light therapy and Alzheimer's disease and related dementia: past, present, and future. J Alzheimers Dis. 2013;33(4):913-22. doi: 10.3233/JAD-2012-121645. PMID 23099814
- [Result] Garin N, Olaya B, Miret M, Ayuso-Mateos JL, Power M, Bucciarelli P, Haro JM. Built environment and elderly population health: a comprehensive literature review. Clin Pract Epidemiol Ment Health. 2014 Oct 21;10:103-15. doi: 10.2174/1745017901410010103. eCollection 2014. PMID 25356084